CLINICAL TRIAL: NCT01062776
Title: New Method to Detect Dehydration
Brief Title: Kinetic Method to Detect Dehydration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sodertalje Hospital (Other)
Responsible Party: Robert Hahn, Södertälje Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: M114-09
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2009-11

CONDITIONS: Dehydration
Keywords: dehydration; fluid therapy; pharmacokinetics; hemoglobin
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5 ml/kg of fluid, no dehydration (Placebo Comparator): Volunteers receive an intravenous infusion of acetated Ringers solution over 15 min without preceding deliberate dehydration with furosemide.
  Interventions: Biological: Placebo
- 10 ml/kg of fluid, no dehydration (Placebo Comparator): Volunteers receive an intravenous infusion of acetated Ringers solution over 15 min without preceding deliberate dehydration with furosemide.
  Interventions: Biological: Placebo
- 5 ml/kg of fluid, dehydration (Experimental): Volunteers receive an intravenous infusion of 5 ml/kg acetated Ringers solution over 15 min after being dehydrated with furosemide.
  Interventions: Biological: Dehydration
- 10 ml/kg of fluid, dehydration (Experimental): Volunteers receive an intravenous infusion of 10 ml/kg acetated Ringers solution over 15 min after being dehydrated with furosemide.
  Interventions: Biological: Dehydration

INTERVENTIONS:
Biological: Dehydration — Furosemide 5 mg is given intravenously over 2 hours until approximately 2 liters of body fluid is lost.
  Other Names: Furosemide för intravenous administration; Acetated Ringer´s solution
  Arms: 10 ml/kg of fluid, dehydration; 5 ml/kg of fluid, dehydration
Biological: Placebo — No dehydration is induced
  Other Names: Acetated Ringer´s solution
  Arms: 10 ml/kg of fluid, no dehydration; 5 ml/kg of fluid, no dehydration

SUMMARY:
1. The distribution and elimination of infusion fluids can be studied by volume kinetics, a mathematical method based on serial analysis of the blood hemoglobin concentration.
2. The hypothesis of the present study is that the elimination of infused fluid is retarded in the presence of dehydration, and that volume kinetics would therefore be capable of detecting dehydration in human subjects.
3. We induce dehydration by injection graded doses of furosemide (a diuretic drug) in healthy volunteers and the kinetics of an infusion of crystalloid fluid is compared to when the same volunteer receives the same fluid without being in a dehydrated state.

DETAILED DESCRIPTION:
1. Fifteen healthy male volunteers are subjected to 4 experiments. They drink 800 ml of water at 6:00 AM to make sure they are not dehydrated when the experiments begin.
2. On two occasions the volunteer receives, at 9:00 AM, an intravenous infusion of acetated Ringer´s solution being either 5 ml/kg or 10 ml/kg, over 15 min. The blood hemoglobin concentration is measured during 16 occasions during 120 min by invasive blood sampling and also non-invasively by a pulse oximeter (Masimo´s Radical 7).
3. On two other occasions, the infusions are preceded for 2 hours of deliberate dehydration. Doses of furosemide 5 mg are repeated 3-4 times with the goal of creating dehydration amounting to approximately 2 liters of fluid. Excreted urine is collected and the volume measured.
4. The kinetics of each infusion is calculated by volume kinetics, and the data compared pairwise from the experiments with and those without dehydration.
5. The accuracy and precision of the non-invasive monitoring of Hgb can be determined.
6. The study is ended with that the Hgb response between the lying and sitting position is compared and with that the fluid balance is restored by ingestion of water.
7. Experiments are performed in the Department of Intensive Care at Linköping University Hospital, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male.

Exclusion Criteria:

* Disease for which daily medication is required.
* Poor peripheral perfusion; defined as a perfusion index, as measured by Masimo´s Radical 7, of 2 or less.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
As determined by volume kinetics, a healthy human male eliminates infused crystalloid fluid more slowly when being in the dehydrated state as compared to when being normohydrated. | December 2010

SECONDARY OUTCOMES:
The volume kinetics of an infusion fluid can/can not be measured as accurately by non-invasive monitoring as by invasive monitoring of the blood hemoglobin concentration | May 2010 (preliminary analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Hahn, MD, PhD, Study Director — Södertälje Hospital
Locations (1):
- Department of Intensive Care, University hospital, Linköping, Sweden, Linköping, Linköping, Sweden

REFERENCES:
- [Derived] Hahn RG, Wuethrich PY, Zdolsek JH. Can perioperative hemodilution be monitored with non-invasive measurement of blood hemoglobin? BMC Anesthesiol. 2021 May 6;21(1):138. doi: 10.1186/s12871-021-01351-4. PMID 33957864